CLINICAL TRIAL: NCT05408338
Title: Acute Effects of Added Sugar Intake on Cerebrovascular Function and Brain Integrity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1718585
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Healthy Diet; Healthy Aging
Keywords: added sugars; brain blood vessel function; brain structure; MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Added Sugar Meal (Experimental): Participants will be provided a meal low in added sugars.
  Interventions: Other: Low Added Sugar Meal
- High Added Sugar Meal (Experimental): Participants will be provided a meal high in added sugars.
  Interventions: Other: High Added Sugar Meal

INTERVENTIONS:
Other: Low Added Sugar Meal — Consumption of a single 1,250 kcal meal containing 16 g of added sugars (5% of total energy)
  Arms: Low Added Sugar Meal
Other: High Added Sugar Meal — Consumption of a single 1,250 kcal meal containing 61 g of added sugars (20% of total energy)
  Arms: High Added Sugar Meal

SUMMARY:
This study will focus on acute effects of added sugars on brain health in a specific age group (30-64 years old). We will provide participants two meals (one meal containing 16 g of added sugars and the other containing 61 g of added sugars) and examine blood vessel function and brain structure using a MRI.

DETAILED DESCRIPTION:
Cardiometabolic risk factors are strongly influenced by lifestyle-related environmental factors including the consumption of an unhealthy Western diet (WD). Added sugars (i.e., caloric sweeteners added to food during processing or preparation) have become a major component of the WD that are especially high in added fructose. Americans currently consume more calories from added sugars than is recommended by the American Heart Association (AHA), leading to an increased risk of cardiovascular disease (CVD), which in turn shares common risk factors with age-related memory loss and dementia. Whereas glucose is used as an immediate energy source or stored as glycogen, fructose is associated with the delayed production of triglycerides (TGs) and uric acid. Previous studies have shown that a single high-sugar meal can increase TGs in the blood 150-180 minutes after meal consumption. Increased blood TGs promote release of harmful substances that contribute to the reduction in blood vessel function and may also impact brain blood vessel function; however, these effects are not well established in humans. Our preliminary data has shown a positive association between high added sugars and plasma TG and uric acid concentration, which has been associated with reduced blood vessel function. However, the direct effects of acute added sugar intake on brain blood vessel function is currently unknown. We have also observed that high blood TGs are associated with reduced microstructural integrity of the hippocampus, a brain structure important for memory and other thinking abilities. Therefore, the purpose of this study is to establish a causal link between high added sugar consumption and reduced brain blood vessel function and microstructural integrity. We propose to examine the acute effects of high TGs and uric acid from a single high-sugar meal on brain blood vessel function and brain integrity. To test this hypothesis, we will conduct a randomized-controlled crossover trial of a high-sugar meal vs. a low-sugar meal. This project has the potential to identify future risk of dementia and other memory-related brain diseases caused from repetitive acute insults from high added sugar consumption and will help us inform the public to make better dietary choices.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent;
* Men and women within the ages of 30-64 years;
* Habitual added sugar intake of <150 kcal/day for men and <100kcal/day for women;
* No allergies/intolerance to ingredients in the study meal (e.g., nuts, gluten)

Exclusion Criteria:

* Blood chemistries indicative of abnormal liver enzymes and renal function;
* Abnormal blood chemistry marker that is +/-2.5x the upper or lower limit;
* Chronic clinical diseases (e.g., coronary artery, peripheral artery, or cerebrovascular diseases, diabetes (type 1 and type 2), stages 5-6 chronic kidney disease, chronic obstructive pulmonary disease);
* Major psychiatric disorder (e.g. schizophrenia, bipolar disorder, major depression within past two years);
* Neurological or autoimmune conditions affecting cognition (e.g. Parkinson's disease, epilepsy, multiple sclerosis, head trauma with loss of consciousness greater than 30 min, large vessel infarct);
* Current medication use likely to affect central nervous system functions (e.g. long active benzodiazepines) and lipid-lowering medications (e.g., statins)
* Conditions which would contra-indicate MRI: implant of pacemakers or pacemaker wires; artificial heart valve; brain aneurysm surgery; middle ear implant; non-removable hearing aid or jewelry; braces; cataract surgery or lens implant; implanted mechanical or electrical device; foreign metallic objects in the body such as bullets, BBs, shrapnel, or metalwork fragments, claustrophobia;
* Current smoking;
* Pregnancy or breastfeeding

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cerebrovascular reactivity at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  % change in total cerebral perfusion measured using pseudo-continuous arterial spin labeling in response to 3-minutes of hypercapnia (+9 mmHg increase in PETCO2)
Change from baseline in hippocampal stiffness after 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Magnetic Resonance Elastography (MRE) of the brain to assess hippocampal viscoelastic properties while the head will be vibrated using the Resoundant acoustic driver system
Change from baseline in hippocampal damping ratio at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Magnetic Resonance Elastography (MRE) of the brain to assess hippocampal viscoelastic properties while the head will be vibrated using the Resoundant acoustic driver system
Change from baseline in uric acid at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Blood biomarker of uric acid (e.g. serum uric acid)
Change from baseline in triglycerides at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Blood biomarker of triglycerides (e.g. serum triglycerides)
Change from baseline in oxidative stress at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Blood biomarker of oxidative stress (e.g. superoxide)

SECONDARY OUTCOMES:
Change from baseline in hippocampal cerebrovascular reactivity at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  % change in total cerebral perfusion measured using pseudo-continuous arterial spin labeling in response to 3-minutes of hypercapnia (+9 mmHg increase in PETCO2)
Changes from baseline in resting cerebral blood flow at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Total cerebral perfusion measured using pseudo-continuous arterial spin labeling
Change from baseline in other lipid profile at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Blood biomarkers of lipid profile (e.g. cholesterol, HDL, LDL, and VLDL)
Change from baseline in blood pressure at 3 hours post-consumption of each meal | Over 2 weeks, at baseline and 3 hours post-consumption of each meal (low and high added sugar), separated by a 1-week washout
  Blood pressure measures at baseline and every half hour until post-consumption of meal

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Martens, PhD, Study Director — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No